CLINICAL TRIAL: NCT00300261
Title: Promoting Self Care Using Telehomecare: Impact on Outcomes
Brief Title: Testing the Effects of Telehealth Monitoring on Rehospitalization and Self Care for Heart Failure Patients in Home Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Kathryn Bowles, van Ameringen Professor in Nursing Excellence, University of Pennsylvania
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 10003907; R01NR008923 (NIH)
Record Dates: First submitted 2006-03-06; First posted 2006-03-08 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2010-03

CONDITIONS: Heart Failure
Keywords: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): receives home care
- 2 (Experimental): receives telehealth monitoring in addition to home care
  Interventions: Behavioral: Telehealth monitoring

INTERVENTIONS:
Behavioral: Telehealth monitoring — Experimental group receives telehealth monitoring equipment in their homes for the duration of home care. Equipment includes blood pressure cuff, scale, and pulse oximeter, or glucometer as needed. Two home care nurses provide video visits with subjects on the days when the home care nurse does not visit. Patients use the equipment daily and the results are downloaded to the nurse's computer at the home care agency where they are checked daily. The nurse acts on any abnormal readings by calling the patient, the home care nurse, or the physician.
  Arms: 2

SUMMARY:
We are testing the use of telehealth technology that includes self monitoring of blood pressure, weight, blood sugar, and oxygen levels for patients with heart failure who are receiving home care. We are interested to learn if using the equipment results in improved self care and decreased incidence of rehospitalization.

DETAILED DESCRIPTION:
Despite telehomecare's potential to enhance patients' self-care in a cost-effective manner, few studies have evaluated its efficacy. Reported studies were conducted prior to the introduction of Medicare's prospective payment system for home care and evaluated the use of telehomecare in addition to traditional home visits. None examined patients' involvement in decision-making regarding the use of such technology in meeting their health care needs. Available data suggest that telehomecare may improve self-care and enhance outcomes for elders with heart failure but major gaps in knowledge exist regarding the clinical and cost effectiveness of this technology when decisions regarding its use are negotiated with patients and when it substitutes for traditional nurse visits under the recently introduced changes in the financing of home health care.

Patient and cost outcomes will include: self-care, health care resource utilization, health status, quality of life, satisfaction, access to care and cost effectiveness. Data analysis will consist of a variety of statistical tests, and estimates of treatment costs. Findings will help guide optimal use of telehomecare in promoting self-care in the growing population of chronically ill elders whose conditions are characterized by high morbidity, complex therapies and poor quality and cost outcomes.

Subjects will be enrolled from the acute care setting and will be randomized to receive home care with or without telehealth monitoring. Baseline and follow-up interviews will be conducted at admission, 60, 120 and 180 days.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of heart failure, English speaking; mentally competent, weigh less than 450 pounds, have a telephone in their home; have Medicare insurance; are able to see, hear, place a cuff on their arm, and stand on a scale to weigh themselves, receiving home care from Penn Care at Home.

Exclusion Criteria:

* cognitive impairment, weight > 450 pounds, receiving disease management or on a heart transplant waiting list, receiving home care from a non- participating agency.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2005-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To learn if using telehealth technology equipment results in improved self care and decreased incidence of rehospitalization. | 60, 120 and 180 days from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn H Bowles, PhD,RN, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States